CLINICAL TRIAL: NCT03650062
Title: Patient-reported Outcome Scale in Acute pancreatitis-an International Prospective Cohort Study
Brief Title: Patient-reported Outcome Scale in Acute Pancreatitis
Acronym: PAN-PROMISE
Status: Completed | Type: Observational
Sponsor: Enrique de-Madaria (Other)
Responsible Party: Sponsor-Investigator, Enrique de-Madaria, Principal Investigator, Hospital General Universitario de Alicante
Organization: Hospital General Universitario de Alicante (Other)
Other Study IDs: PI2016/69
Record Dates: First submitted 2018-08-20; First posted 2018-08-28 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Acute Pancreatitis
Keywords: Patient Reported Outcome Measures; Follow-Up Studies; Patient Outcome Assessment; Treatment Outcome; Pancreatitis, Acute Necrotizing
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PAN-PROMISE study (PAtieNt-rePoRted OutcoMe scale in acute pancreatItis-an international proSpEctive cohort study) aims to measure an outcome variable in acute pancreatitis (AP) based in the patient´s experience. PAN-PROMISE is a cohort study involving patients with AP. The patient´s symptom perception will be compared with the opinion of the clinicians and with clinical outcomes.

DETAILED DESCRIPTION:
Currently, the most important outcome variables in Acute Pancreatitis (AP) are persistent organ failure (POF) and mortality, according to the physician point of view. These variables occur infrequently (<10 and <5% respectively) (Sternby et all, see "References"), therefore, studies designed to assess the effectiveness of new treatments for AP to decrease POF or mortality require a very large sample of patients, which is unfeasible. Currently, clinical trials addressing the management of AP do not take into account Patient Reported Outcome Measures.

PROMS (Patient Reported Outcome Measures) have been defined as any report of the status of a patient's health condition that comes directly from the patient, without interpretation of the patient's response by a clinician or anyone else (first link in "References"). PROMS are gaining importance as a tool to design outcome variables. This kind of measurement has been recently included in the quality assesment approaches (Crossing the Quality Chasm: A New Health System for the 21st Century, see "References"), being PROMS a useful tool to improve the triple aim framework of better quality, appropriate utilization, and enhanced patient experience (second link in "References"). The aim of PAN-PROMISE is to incorporate an outcome variable in AP based in the patient´s experience. For this purpose the investigators involved in this project have developed a new instrument based on symptoms found to be important for the patient. This new instrument is intended to be a simple quantitative variable, relevant for the patient, that can be useful to test new treatments for AP without the need for a very large sample size, fulfilling the requirements of the triple aim framework by incorporating an outcome measurement defined by the patient.

Hypothesis:

* PROMS must be incorporated to patient care and research in AP to improve the triple aim framework of better quality, appropriate utilization, and enhanced patient experience
* A PROMS scale is a useful outcome variable to investigate new treatments in AP
* The different severity categories of the revision of the Atlanta Classification (RAC) have different scores on the PROMS scale in acute pancreatitis: severe greater than moderate and mild, moderate greater than mild.
* Increasing scores on the PROMS scale are associated to increased morbidity

Aims:

* Main aim 1: to measure patient´s symptoms during an episode of AP and to correlate the intensity of these symptoms to clinical outcomes
* Main aim 2: to design and validate a PROMS scale in AP intended to be an suitable outcome variable in future trials addressing the management of AP

Methods

Part 1: development of the PAN-PROMISE instrument The PAN-PROMISE research team developed a qualitative study in which three nominal groups were conducted, two with patients who had suffered an acute pancreatitis (AP) in hospitals in Alicante (Universitarian General Hospital)), and Valencia (Clinic Hospital), Spain and another with clinicians from the Alicante region with experience in treating patients with AP. Participants were asked about the symptoms that cause the most discomfort and concern to patients at three specific times: before receiving treatment for AP, during hospital admission and after discharge. The perspectives of patients and professionals were compared. From the information gathered in the nominal groups, a first version of a PROMS questionnaire was elaborated and shared with an international group of gastroenterologists, experienced in the management of pancreatitis, from 4 countries (Germany, Spain, USA, India and Turkey) through an online application to determine to what extent these experiences were shared in frequency and intensity by patients in these different countries. With all this information, a PROMS instrument was generated.

Part 2: measurement of patient´s symptoms in an international cohort study

2.1 Design. The PAN-PROMISE instrument is being measured in patients participating in a multicenter international prospective cohort study. Consecutive adult patients with AP are eligible after signed informed consent.

2.2 Center recruitment The PAN-PROMISE study has been endorsed by the Spanish Association of Pancreatology (AESPANC), the Spanish Association of Gastroenterology (AEG) and the International Association of Pancreatology (IAP); these associations shared the project with their members and through their social networks, calling for researchers and centers to join this initiative. PAN-PROMISE has also a webpage www.promisepancreatitis.com to promote center recruitment.

2.3 Patient registry PAN-PROMISE measurement will rely on a patient registry hosted in the Spanish Association of Gastroenterology (AEG) REDCap node. AEG offered this REDCap web-based online patient registry tool at no cost. Claudia Sánchez-Marin, a gastroenterologist, is on charge of quality control (data validation, data checks, contact with researchers to solve issues). The REDCap online registry was designed with logical rules to ensure good quality data entry, including mandatory fields to enter, logical ranges for quantitative variables, alarms if logical rules are not coherent (for example to have persistent organ failure but to classify the episode as mild or moderate), expanding fields only available in the presence of certain circumstances (for example, detailed organ failure description is only available if the patient had organ failure).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 and <80 years.
* Karnofsky performance status previous to AP 100 (normal, no complaints, no evidence of disease), 90 (able to carry on normal activity; minor signs or symptoms of disease) or 80 (normal activity with effort; some signs or symptoms of disease).
* Acute pancreatitis defined as at least 2 of the following 3 criteria: A) Typical abdominal pain, B) Elevation of amylase and/or lipase more than 3 times the upper limit of normality, and C) Imaging (preferably CT and/or MR) compatible with AP.
* Written informed consent.

Exclusion Criteria:

* Time between onset of symptoms and presentation in the emergency room (ER) greater than 48 hours (we do not consider as onset of symptoms previous self-limited heraldic biliary pain)
* Recruitment >24h after presentation in the ER
* Karnofsky performance status previous to AP 70 (Cares for self; unable to carry on normal activity or to do active work) or less
* Inability to express or understand the instructions of the study (severe congenital or acquired intellectual deficit).
* More than 1 previous episode of AP.
* Chronic pancreatitis.
* Presence of diseases or conditions different from AP that may interfere with the scale: other causes of abdominal pain (especially acute cholecystitis; Note: choledocholithiasis-acute cholangitis is not an exclusion criteria), obstruction of the digestive tract (peptic pyloric stenosis, gastrointestinal anastomotic stenosis, diabetic gastroparesis, gastrointestinal neoplasia...), nausea-vomiting (brain tumor, chemotherapy...) or weakness (pre-existing anemia with Hb <9 mg/dL, heart failure or respiratory insufficiency associated with minimal effort dyspnea, or domiciliary treatment with O2, advanced neoplasms or other debilitating diseases).

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted with acute pancreatitis in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-03 (Actual)

PRIMARY OUTCOMES:
Severity of acute pancreatitis according to the revised Atlanta classification [incidence of local and/or systemic complications] | Up to 15 days after hospital discharge from index hospital admission
  Mild acute pancreatitis (no complications), moderately severe acute pancreatitis (local complications and/or transient (≤48h) organ failure and/or exacerbation of previous comorbidity), severe acute pancreatitis (persistent (>48h) organ failure) (see revised Atlanta classification, Banks et al, Gut 2013)
PAN-PROMISE patient reported outcome measurement instrument | From within 24h after admission to 15 days after discharge
  PROMISE SCALE (Patient-reported Outcome Scale in Acute pancreatitis) Each item is scored from 0 to 10 ( worst score in the last 24h): 0 none, 10: the highest possible intensity according to the patient
  1. Pain, especially in the abdomen, chest or back
  2. Abdominal distention (bloating, sensation of excess gas)
  3. Difficulty eating, sensation of food being stuck in the stomach
  4. Difficulty with bowel movements (constipation or straining on bowel movements)
  5. Nausea and/or vomiting
  6. Thirst
  7. Weakness, lack of energy, fatigue, difficulty moving

SECONDARY OUTCOMES:
EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30) Version 3.0 | 15 days after hospital discharge
  EORTC QLQ-C30, a widely used and validated quality of life scale, includes 28 questions with a four-point scale: "Not at all" (1 point), "A little" (2), "Quite a bit" (3) and "Very much." (4); 4 means an important impact on quality of life. The last 2 questions are scored from 1 (very poor) to 7 (excellent), being 7 indicative of excellent quality of life.
C-reactive protein | 48 and 72h after recruitment
  A marker of inflammation
Local complications (incidence of pancreatic/peripancreatic necrosis and acute peripancreatic fluid collections) | Up to 15 days after hospital discharge from index hospital admission
  Defined according to the revised Atlanta classification (Banks et al, Gut 2013)
Need for invasive treatment | Up to 15 days after hospital discharge from index hospital admission
  Endoscopic, percutaneous or surgical drainage or necrosectomy
Need for nutritional support | Up to 15 days after hospital discharge from index hospital admission
  Need for enteral and/or parenteral nutritional support
Admission in the Intensive Care Unit | Up to 15 days after hospital discharge from index hospital admission
  Need for intensive care support
Hospital stay | Up to 15 days after hospital discharge from index hospital admission
  Days, on index admission
Organ failure | Up to 15 days after hospital discharge from index hospital admission
  Transient and persistent organ failure defined according to the revised Atlanta classification (Banks et al, Gut 2013)
Mortality | Up to 15 days after hospital discharge from index hospital admission
  Mortality during index admission
Hospital readmission | Up to 15 days after hospital discharge from index hospital admission
  Hospital readmission due to symptom relapse or complications of index acute pancreatitis
Systemic Inflammatory Response Syndrome (SIRS) | Up to 15 days after hospital discharge from index hospital admission
  Presence of SIRS and persistent (>48h) SIRS

CONTACTS AND LOCATIONS:
Overall Officials: José Joaquín Mira, PsyD PhD, Study Director — Universidad Miguel Hernandez de Elche; Enrique de-Madaria, MD PhD, Principal Investigator — Hospital General Universitario de Alicante
Locations (26):
- Johns Hopkins Medical Center, Baltimore, Maryland, United States
- Hospital Universitario San Ignacio, Bogotá, Colombia
- Attikon University Hospital, Athens, Greece
- Hungary (2):
  - Centre for Translational Medicine, University of Pécs, Pécs
  - University of Szeged, Szeged
- Dip.Medicina-Università degli Studi di Verona, Verona, Italy
- Vilnius University, Vilnius, Lithuania
- Servicio de Cirugía General, IMSS, León, Guanajuato City, Mexico
- Medical University of Łódź, Lodz, Poland
- Portugal (2):
  - Fernando Fonseca Hospital, Amadora
  - Centro Hospitalar Tondela-Viseu, Viseu
- Romania (2):
  - Emergency Hospital of Bucharest, Bucharest
  - Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca
- Immanuel Kant Baltic Federal University, Kaliningrad, Russia
- Konkuk University School of Medicine, Seoul, South Korea
- Spain (10):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Santa María, Lleida
  - Hospital San Pedro, Logroño
  - Hospital Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
- Medical Institute Lviv, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
The whole database will be offered to the study collaborators who actively recruited patients
Time Frame: The database will be available after publication of the PAN-PROMISE study
Access Criteria: Collaborating researchers who recruited patients will be able to apply for access to the database. The protocol of the proposed study will be considered by the PAN-PROMISE scientific committee

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Result] Sternby H, Bolado F, Canaval-Zuleta HJ, Marra-Lopez C, Hernando-Alonso AI, Del-Val-Antonana A, Garcia-Rayado G, Rivera-Irigoin R, Grau-Garcia FJ, Oms L, Millastre-Bocos J, Pascual-Moreno I, Martinez-Ares D, Rodriguez-Oballe JA, Lopez-Serrano A, Ruiz-Rebollo ML, Viejo-Almanzor A, Gonzalez-de-la-Higuera B, Orive-Calzada A, Gomez-Anta I, Pamies-Guilabert J, Fernandez-Gutierrez-Del-Alamo F, Iranzo-Gonzalez-Cruz I, Perez-Munante ME, Esteba MD, Pardillos-Tome A, Zapater P, de-Madaria E. Determinants of Severity in Acute Pancreatitis: A Nation-wide Multicenter Prospective Cohort Study. Ann Surg. 2019 Aug;270(2):348-355. doi: 10.1097/SLA.0000000000002766. PMID 29672416
- [Derived] de-Madaria E, Sanchez-Marin C, Carrillo I, Vege SS, Chooklin S, Bilyak A, Mejuto R, Mauriz V, Hegyi P, Marta K, Kamal A, Lauret-Brana E, Barbu ST, Nunes V, Ruiz-Rebollo ML, Garcia-Rayado G, Lozada-Hernandez EE, Pereira J, Negoi I, Espina S, Hollenbach M, Litvin A, Bolado-Concejo F, Vargas RD, Pascual-Moreno I, Singh VK, Mira JJ. Design and validation of a patient-reported outcome measure scale in acute pancreatitis: the PAN-PROMISE study. Gut. 2021 Jan;70(1):139-147. doi: 10.1136/gutjnl-2020-320729. Epub 2020 Apr 3. PMID 32245906
- See also: Guidance for Industry Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims — https://www.fda.gov/downloads/drugs/guidances/ucm193282.pdf
- See also: Institute for Healthcare Improvement (IHI): The IHI Triple Aim — http://www.ihi.org/Engage/Initiatives/TripleAim/Pages/default.aspx